CLINICAL TRIAL: NCT02095990
Title: Efficacy and Safety of a 4% Hydroquinone Cream (Melanoderm 4%) for the Treatment of Melasma: a Randomized Controlled Split-face Study
Brief Title: Efficacy and Safety of a 4% Hydroquinone Cream for the Treatment of Melasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECM2013
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2015-04

CONDITIONS: Facial Melasma
Keywords: Facial Melasma
MeSH Terms: interventions — hydroquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroquinone (Experimental): Hydroquinone 4% Cream will be applied in one side of the face while the other side of the face receives placebo.
  Half of the patients will receive Hydroquinone on the right side of the face and the other half on the left side.
  It will be applied daily, at night, during 8 weeks.
  Interventions: Drug: Hydroquinone
- Placebo (Placebo Comparator): Placebo cream (vehicle of Hydroquinone 4% cream), will be applied in one side of the face, while the other side receives the active treatment.
  Half of the patients will receive Hydroquinone on the right side of the face and the other half on the left side.
  It will be applied daily, at night, during 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroquinone
  Arms: Hydroquinone
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the ability of a new 4% Hydroquinone formulation (Melanoderm 4% Crema) to reduce melasma on the face, using a split-face randomization design, evaluating the MASI Score from baseline to week 4 and week 8, in both half-faces receiving active treatment vs. placebo.

To assess the tolerance of a new 4% Hydroquinone formulation (Melanoderm 4% Crema) on the face.

To assess patients' satisfaction regarding Melanoderm 4% Crema after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged between 18-65 years old.
* Fitzpatrick phototypes I to IV.
* Presenting moderate to severe facial melasma facial, with a basal Melasma Area and Severity Index (MASI Index) between 10 and 20.
* Women of childbearing potential must use an adequate contraceptive method to avoid pregnancy and must have a negative pregnancy test in a maximum of 72 hours before receiving the trial treatment.
* Breastfeeding women will not be included in the study.
* Having given freely and expressly her informed consent.

Exclusion Criteria:

* Those with any history of allergy or hypersensitivity to a cosmetic product, hydroquinone, or one of the ingredients of the investigational products.
* Fitzpatrick phototype V.
* Skin pigmentation diseases different to melasma.
* Evidence of active cancer disease or diagnosis of cancer in the last year.
* Those receiving any topical or oral treatment that could interfere with melasma.
* Pregnant or breastfeeding women, or those expecting to get pregnant during the study.
* Evidence or suspicion of low compliance with the study visits and procedures.
* Participation in other clinical trial simultaneously or in the previous 3 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To assess the ability of a new 4% Hydroquinone formulation (Melanoderm 4% Crema) to reduce melasma on the face. | Baseline, week 4, week 8.
  Efficacy assessments will be measured by the Melasma Area and Severity Index (MASI Index) at baseline, week 4 and week 8 (end of treatment).

SECONDARY OUTCOMES:
To assess the tolerance of a new 4% Hydroquinone formulation (Melanoderm 4% Crema) on the face. | Week 4, Week 8, Follow-up period (Week 12)
  Adverse events will be recorded throughout the study and 30 days after the end of treatment.

OTHER OUTCOMES:
To assess patients' satisfaction regarding Melanoderm 4% Crema. | Week 8
  Patients' satisfaction in terms of efficacy and safety will be evaluated by a Visual Analogic Scale at week 8, which will be completed for each side of the face independently.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Puig, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain